CLINICAL TRIAL: NCT05287100
Title: To Assess the Efficacy of Midodrine in Prevention of Cirrhosis Related Complications in Children Awaiting Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-49
Record Dates: First submitted 2022-03-11; First posted 2022-03-18 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis | interventions — Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midodrine (Experimental): Midodrine starting at 0.25mg/kg/day in 2-3 divided doses, increased to 0.5mg/kg/day after 7 days if MAP does not increase by >10% ; Midodrine dosage will be decreased by 25% in case of arterial hypertension (>95th centile BP for the age). Also Standard medical therapy as per departmental protocol will be continued
  Interventions: Drug: Midodrine Oral Tablet; Other: Standard Medical Treatment
- Standard medical therapy (Active Comparator): Standard medical therapy as per departmental protocol
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Drug: Midodrine Oral Tablet — Midodrine starting at 0.25mg/kg/day in 2-3 divided doses, increased to 0.5mg/kg/day after 7 days if MAP does not increase by >10% ; Midodrine dosage will be decreased by 25% in case of arterial hypertension (>95th centile BP for the age). Also Standard medical therapy as per departmental protocol will be continued
  Arms: Midodrine
Other: Standard Medical Treatment — Albumin infusion 1g/kg/day - maximum 20gm/day and repeat till serum albumin reaches 2.8g/dl If serum albumin is < 2.8g/dl SBP - Day 1 and Day 3
  For Ascites :
  Restriction of sodium to < 2meq/kg/day A combination of a distal-acting diuretic (spironolactone, 3-6 mg/ kg/day) and loop-acting diuretic (furosemide,0.5- 2 mg/kg per day) was given with dose escalation by one step at a time if there is no decrease in weight (by ≥ 0.5 %/day) after 5-7 days Therapeutic paracentesis (>50ml/kg) with infusion of albumin (8 g/L) performed for tense, symptomatic ascites
  For Spontaneous Bacterial Peritonitis :
  IV antibiotics for 7 days Albumin Infusion on Day 1 and Day 3

SUMMARY:
Children with cirrhosis awaiting transplantation are more proned to develop various complications. The pathogenesis of cirrhotic complications (ascites, hyponatremia, acute kidney injury) includes release of vasodilatory molecules like nitric oxide, damage associated molecular pathogens (DAMPs) and pattern associated molecular pathogens (PAMPs) secondary to bacterial translocation, which causes splanchnic bed vasodilation resulting in activation of renin-angiotensin and aldosterone axis(RAAS) causing sodium and water retention and renal vasoconstriction [1].

The development of complications in these children may result in death or may preclude them from reaching upto liver transplantation [2].

Midodrine is an α1 adrenergic receptor agonist, which increases vascular tone causing rise in the blood pressure, thereby improving renal perfusion and causes RAAS deactivation. The effects of midodrine is documented in reduction of refractory ascites, hepatorenal syndrome and hyponatremia[2-4].

One group will receive only standard medical therapy and other group will receive midodrine and standard medical therapy for 6 months. Mean arterial pressure will be monitored at every OPD visit. At the end of 12 weeks, and 24 weeks, plasma renin activity, incidence of complications related to cirrhosis like new onset ascites, increase in grade of ascites, hyponatremia, acute kidney injury and spontaneous bacterial peritonitis will be assessed. Also the transplant free survival and need for albumin transfusion will be compared between the two groups.

In case of liver transplantation or death before 6 months, midodrine will be stopped

DETAILED DESCRIPTION:
Aim: To determine the efficacy of midodrine in preventing development of complications in children with cirrhosis awaiting liver transplantation

Primary Objective:

1) To compare incidence of complications (Acute kidney injury, New onset ascites or increase in grade of ascites, Spontaneous bacterial peritonitis, Hyponatremia, Hepatic encephalopathy) of cirrhosis in patients receiving midodrine (at a dose of 0.25 - 0.5mg/kg/day) and standard medical therapy versus standard medical therapy alone for 6 months

Secondary Objectives:

* Frequency of development of new onset ascites or increase in grade of ascites by 6 months
* Change in serum sodium from baseline to 6 months
* Change in Mean arterial pressure (MAP) at 1 week and then 2 weekly till the end of the study
* Plasma renin activity at baseline, at 12 weeks and 24 weeks
* Frequency of development of SBP over 6 months
* Change in eGFR from baseline to 6 months
* Frequency of developing AKI by 6 months
* Frequency of development of Hepatic encephalopathy by 6 months
* Proportion of patients developing hypertension at 6 months
* Frequency of development of drug related adverse effects by 6 months
* Requirement of albumin infusion in 2 groups
* Transplant free survival

Methodology:

* Study population :Children and Adolescents of age group upto 18 years with cirrhosis and PELD/ MELDNa score more than 14, on waitlist for liver transplantation following up in the Pediatric Hepatology Department
* Study design: Open label RCT (computer based randomization - block randomization with block size of 4)
* Study period: 6 months weeks for each patient; The study will be conducted between January 2022 and July 2023
* Sample size:
* Pilot study - 10 patients in each group

ELIGIBILITY:
Inclusion Criteria:

Children and Adolescents of age group upto 18 years with cirrhosis and PELD/ MELDNa score more than 14, on waitlist for liver transplantation following up in the Pediatric Hepatology Department, ILBS will be prospectively included in this study after informed consent

Exclusion Criteria:

Presence of Portal vein thrombosis Renal or cardiovascular disease or arterial hypertension Presence of HCC

Ages: 10 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Complications between the two groups | 6 months
  • To compare incidence of complications (Acute kidney injury, New onset ascites or increase in grade of ascites, Spontaneous bacterial peritonitis, Hyponatremia, Hepatic encephalopathy) of cirrhosis in patients receiving midodrine (at a dose of 0.25 - 0.5mg/kg/day) and standard medical therapy versus standard medical therapy alone for 6 months

SECONDARY OUTCOMES:
• Frequency of development of new onset ascites or increase in grade of ascites by 6 months | 6 months
Change in serum sodium from baseline to 6 months | 6 months
Change in Mean arterial pressure (MAP) at 1 week and then 2 weekly till the end of the study | 6 months
Plasma renin activity at baseline, at 12 weeks and 24 weeks | 6 months
Frequency of development of SBP over 6 months | 6 months
Change in eGFR from baseline to 6 months | 6 months
Frequency of developing AKI by 6 months | 6 months
Frequency of development of Hepatic encephalopathy by 6 months | 6 months
Proportion of patients developing hypertension at 6 months | 6 months
Frequency of development of drug related adverse effects by 6 months | 6 months
Requirement of albumin infusion in 2 groups | 6 months
Transplant free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Seema Alam, MD, Study Director — ILBS
Locations (1):
- Institute of liver and biliary sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashritha A, Lal BB, Khanna R, Sood V, Sood AK, Alam S. Midodrine reduces new-onset acute kidney injury and hyponatremia in children with cirrhosis and ascites awaiting liver transplantation: Results from an open-label RCT. J Pediatr Gastroenterol Nutr. 2024 Feb;78(2):350-359. doi: 10.1002/jpn3.12077. Epub 2023 Dec 11. PMID 38374552